CLINICAL TRIAL: NCT01556334
Title: Preterm Premature Rupture of Membranes: Erythromycin Versus Azithromycin a Randomized Trial Comparing Their Efficacy to Prolong Latency (PEACE Trial)
Brief Title: Erythromycin Versus Azithromycin in Preterm Premature Rupture of Membranes
Acronym: PEACE
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated before starting due to need for IND determined by FDA.
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: PEACE Trial-1011004323
Record Dates: First submitted 2012-03-14; First posted 2012-03-16 (Estimated); Last update posted 2024-10-15 (Actual); Status verified 2014-03

CONDITIONS: Preterm Premature Ruptured Membranes
Keywords: premature ruptured membranes; azithromycin; erythromycin; latency; antibiotics
MeSH Terms: interventions — Azithromycin; Erythromycin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azithromycin (Experimental): Azithromycin 1g po
  Interventions: Drug: Azithromycin
- Erythromycin (Active Comparator): Erythromycin IV followed by po for a total of 5 days.
  Interventions: Drug: Erythromycin

INTERVENTIONS:
Drug: Azithromycin — Azithromycin 1g po
  Other Names: amp/azithro
  Arms: Azithromycin
Drug: Erythromycin — Erythromycin IV then PO
  Other Names: amp/erythro
  Arms: Erythromycin

SUMMARY:
Preterm Premature Rupture of Membranes (PPROM) is treated with an antibiotic, erythromycin or azithromycin, to prolong pregnancy. Erythromycin is taken for several days and can result in stomach upset in some patients, causing them to stop taking the medication. Therefore, azithromycin is often prescribed instead. Azithromycin is usually taken only once and stomach upset is not seen or greatly reduced. The goal of this study is to see if there is a difference between the antibiotic (azithromycin) compared to the antibiotic (erythromycin) in prolonging pregnancy in patients with Preterm Premature Rupture of Membranes (PPROM). The working hypothesis is that there is no difference in the clinical effectiveness between antibiotic regimens containing the macrolides azithromycin and erythromycin for prolonging latency in PPROM.

DETAILED DESCRIPTION:
Preterm, premature rupture of membranes complicates 140,000 pregnancies annually in the United States and is a major contributor to pre-term births and resultant neonatal morbidity and mortality. Typically, a brief period of latency exists after PPROM, with 70-80% of women delivering within the 1st week of membrane rupture. It has been shown through numerous well-conducted trials that antibiotics can prolong this latency time to delivery. Mercer and et al., demonstrated that the administration of ampicillin with erythromycin prolonged the median time to delivery, in comparison to placebo, from 2.9 to 6.1 days. This regimen has now become the standard protocol of treatment in PPROM patients. However, this protocol requires a multi-day dosing regimen of erythromycin and it has been known to have untoward gastrointestinal side effects leading to decreased patient compliance. To overcome these challenges, azithromycin, a newer 2nd generation macrolide, is now commonly being used as a substitution on many of our labor and delivery units nationwide. Azithromycin has a long intracellular half-life, which allows for a more patient friendly one-time dosing regimen; in addition many of the unwanted side effects seen with erythromycin are not seen or greatly reduced with azithromycin, making it an attractive alternative. Despite its popular use, there is a lack of evidence in the literature to support azithromycin as an agent to prolong latency. The purpose of this study is to demonstrate that there is no difference in the clinical effectiveness of azithromycin and erythromycin for prolonging latency in PPROM patients. This trial will be a prospective randomized trial performed in singleton pregnancies with PPROM between 24 0/7 - 32 0/7 weeks gestation. The protocol will enroll 250 eligible women who will then be randomized to receive either azithromycin 1 gm orally at enrollment or erythromycin 250mg IV every 6 hours for 48 hours followed by 500mg orally every 8hours for 5 days. All women will also receive the standard ampicillin 2gm IV every 6 hours followed by amoxicillin 250mg orally every 8 hours for 5 days. The primary outcome measure is the time of latency between the two groups. Secondary outcomes of neonatal death, need for oxygen supplementation, ventilation, and neonatal infection, will also be reviewed. In addition, side effect profiles between the two will be assessed in a post treatment patient survey.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at least 18 years old
* Gestational age of 24 0/7 to 32 0/7 weeks
* Singleton gestation
* Randomization within 36 hours of rupture of membranes.
* Cervical dilation less than or equal to 4 cm.

Exclusion Criteria:

* Known lethal fetal anomaly
* Vaginal bleeding not associated with labor
* Maternal or fetal indication for delivery
* Diagnosis of chorioamnionitis on admission
* Cervical cerclage in place
* Placenta previa or other known placental anomalies
* Use of antibiotic therapy within 5 days.
* Allergy or other contraindications to erythromycin/azithromycin or steroid use.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Time to delivery | 2 years
  To compare the mean time to delivery, using azithromycin versus erythromycin to prolong latency in PPROM patients. The working hypothesis for this aim is that there is no difference in the clinical effectiveness between antibiotic regimens containing the macrolides azithromycin and erythromycin for prolonging latency in PPROM.

CONTACTS AND LOCATIONS:
Overall Officials: David M Haas, MD, MS, Principal Investigator — IU School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States